CLINICAL TRIAL: NCT07238296
Title: Prophylactic Endoscopic Sphincterotomy in Patients Unfit for Cholecystectomy After an Acute Biliary Pancreatitis Episode - an Open-label, Two-armed, Randomized Controlled Trial
Brief Title: Prophylactic Sphincterotomy in Acute Biliary Pancreatitis Patients Unfit for Surgery
Acronym: PROSECCO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NNGYK/34436-6/2025
Record Dates: First submitted 2025-09-22; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Acute Biliary Pancreatitis
Keywords: ERCP; prophylactic sphincterotomy; cholecystectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic endoscopic sphincterotomy (Active Comparator): Papillary cannulation and sphincterotomy techniques will be performed in adherence to the recommendations outlined in the ESGE (European Society of Gastrointestinal Endoscopy) guideline. All recommended measures for post-ERCP (Endoscopic Retrograde Cholangiopancreatography) pancreatitis prevention must be implemented, including the use of prophylactic pancreatic stents, rectal nonsteroidal anti-inflammatory drugs, and optimal hydration protocols where appropriate.
  All rescue techniques may be utilized if necessary, in accordance with clinical judgment and guideline recommendations.
  ERCP/ES (endoscopic sphincterotomy) will be performed by an experienced endoscopist, defined as someone who has performed more than 300 ERCPs in their lifetime and maintains a native papilla cannulation success rate of at least 90%.
  If the ES cannot be performed during the initial ERCP, the number of further attempts is under the discretion of the endoscopist.
  Interventions: Procedure: Prophylactic endoscopic sphincterotomy
- Conservative treatment (No Intervention): This study arm will follow a conservative treatment strategy, and no endoscopic procedures will be performed.

INTERVENTIONS:
Procedure: Prophylactic endoscopic sphincterotomy — Participants in this arm will undergo prophylactic endoscopic sphincterotomy performed by experienced endoscopists, with all recommended preventive measures against post-endoscopic retrograde cholangiopancreatography pancreatitis (PEP) applied according to international guidelines.
  Arms: Prophylactic endoscopic sphincterotomy

SUMMARY:
This is a prospective, multicenter, open-label, randomized controlled trial designed to evaluate the efficacy and safety of prophylactic endoscopic sphincterotomy (ES) in frail patients unfit for cholecystectomy following an episode of acute biliary pancreatitis (ABP).

Eligible patients will be randomized in a 1:1 ratio to either prophylactic ES during the index admission or conservative treatment. The primary endpoint is a composite of recurrent pancreatobiliary events within 12 months, including recurrent ABP, cholangitis, choledocholithiasis requiring endoscopic retrograde cholangiopancreatography (ERCP), or cholangiogenic liver abscess. Secondary outcomes include mortality, pancreatobiliary events requiring intensive care unit admission, post-ERCP complications, cholecystitis, and length of hospitalization.

A total of 92 patients will be enrolled. The trial will be led by the Institute of Pancreatic Diseases, Semmelweis University, Budapest, Hungary, and conducted in accordance with Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (above 18 years)
2. naïve papilla
3. evidence of AP based on the Atlanta criteria:

   * pain in the upper abdomen
   * serum amylase or lipase concentration > 3 times the upper limit of normal
   * imaging features of acute pancreatitis on abdominal imaging
4. high probability of a biliary etiology:

   * gallstones or biliary sludge on imaging (any type)
   * dilated common bile duct on imaging defined as > 8 mm in patients ≤ 75 years or > 10 mm in patients > 75 years
   * abnormal liver enzymes (alanine aminotransferase [ALT] two times the upper limit of normal)
5. patients unfit for surgery due to the attending physician's decision e.g. American Society of Anesthesiologists (ASA) class ≥ III; severe heart failure with reduced ejection fraction <40%, severe uncontrolled hypertension, chronic kidney disease stage four or five

Exclusion Criteria:

1. previous cholecystectomy
2. previous endoscopic sphincterotomy or pancreatobiliary stenting
3. ERCP/ES is recommended by the guidelines (3)

   * sign of cholangitis
   * presence of CBD stone on any imaging
   * signs of stone in endoscopic ultrasonography or magnetic resonance imaging in case of abnormal liver enzymes (persistently elevated ALT and aspartate aminotransferase (AST) with less than a 20% decrease over four days) or dilated CBD (defined as above)
4. chronic pancreatitis
5. estimated life expectancy < 12 months
6. ERCP is contraindicated, e.g. the procedure cannot be carried out safely due to the patient's comorbidities or physical status; high risk of bleeding or contraindication of the discontinuation of the anticoagulation therapy.
7. ERCP is technically not feasible due to altered anatomy, e.g., total gastrectomy, Roux-en-Y gastric bypass anatomy
8. pancreatobiliary malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Recurrent pancreatobiliary events | 1 year
  Composite endpoint:
  * cholangitis - Tokyo guidelines
  * recurrent acute biliary pancreatitis - revised Atlanta criteria
  * choledocholithiasis - imaging/ERCP confirmation
  * cholangiogenic liver abscess - imaging plus clinical diagnosis

SECONDARY OUTCOMES:
Number of participants with recurrent acute biliary pancreatitis, cholangitis, choledocholithiasis, or cholangiogenic liver abscess (individual components of the composite primary outcome) | At 3, 6, 9, and 12 months.
  Each component event will be reported separately as the number of participants experiencing the event during follow-up. Definitions: recurrent acute biliary pancreatitis (revised Atlanta criteria), cholangitis (Tokyo guidelines), choledocholithiasis (imaging/ERCP-confirmed bile duct stone), cholangiogenic liver abscess (imaging and clinical diagnosis).
Length of hospitalization | From enrollment to one month.
  The number of days from hospital admission until discharge, as determined by the treating physician based on clinical stability and institutional criteria. Results will be reported as days of hospitalization per participant, summarized using descriptive statistics (mean, median, interquartile range and standard deviation).
Pancreatobiliary events requiring intensive care unit admission | At 3, 6, 9, and 12 months.
  Number of pancreatobiliary events (recurrent acute biliary pancreatitis, cholangitis, choledocholithiasis, cholangiogenic liver abscess) resulting in intensive care unit admission. Events will be defined according to standard criteria (revised Atlanta criteria for pancreatitis, Tokyo guidelines for cholangitis, imaging/ERCP confirmation for choledocholithiasis, and imaging plus clinical diagnosis for liver abscess).
Mortality associated with pancreatobiliary events | At 3, 6, 9, and 12 months.
  Deaths directly attributable to pancreatobiliary events (recurrent acute biliary pancreatitis, cholangitis, choledocholithiasis, cholangiogenic liver abscess), adjudicated by the study committee. Events will be defined according to standard criteria (revised Atlanta criteria for pancreatitis, Tokyo guidelines for cholangitis, imaging/ERCP confirmation for choledocholithiasis, and imaging plus clinical diagnosis for liver abscess).
All-cause mortality | At 3, 6, 9, and 12 months.
  Death from any cause during follow-up.
Acute cholecystitis | At 3, 6, 9, and 12 months.
  Incidence of acute cholecystitis (Tokyo Guidelines).
Post-endoscopic retrograde cholangiopancreatography pancreatitis | Peri-procedural.
  Incidence of pancreatitis (revised Atlanta-criteria) following endoscopic retrograde cholangiopancreatography, with focus on moderate and severe cases
Other endoscopic retrograde cholangiopancreatography-related complications | Peri-procedural.
  Incidence of adverse events related to endoscopic retrograde cholangiopancreatography, including bleeding, cholangitis, and perforation.
  Complications will be defined according to clinical, laboratory, endoscopic, and imaging findings, and classified by severity based on the need for intervention, hospitalization, or prolonged recovery.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be available upon reasonable request to the study investigators after publication.
Supporting Information: Study Protocol, SAP
Time Frame: It will be available from 6 months after publication of the primary results and will remain available for at least 5 years thereafter.
Access Criteria: Researchers with a methodologically sound proposal may request access to the de-identified IPD. Requests should be submitted to the corresponding author. Data will be shared after approval of the request and signing a data-sharing agreement, through secure institutional data transfer.

REFERENCES:
- [Background] Hajibandeh S, Jurdon R, Heaton E, Hajibandeh S, O'Reilly D. The risk of recurrent pancreatitis after first episode of acute pancreatitis in relation to etiology and severity of disease: A systematic review, meta-analysis and meta-regression analysis. J Gastroenterol Hepatol. 2023 Oct;38(10):1718-1733. doi: 10.1111/jgh.16264. Epub 2023 Jun 27. PMID 37366550
- [Background] Dedemadi G, Nikolopoulos M, Kalaitzopoulos I, Sgourakis G. Management of patients after recovering from acute severe biliary pancreatitis. World J Gastroenterol. 2016 Sep 14;22(34):7708-17. doi: 10.3748/wjg.v22.i34.7708. PMID 27678352
- [Background] Testoni PA, Mariani A, Aabakken L, Arvanitakis M, Bories E, Costamagna G, Deviere J, Dinis-Ribeiro M, Dumonceau JM, Giovannini M, Gyokeres T, Hafner M, Halttunen J, Hassan C, Lopes L, Papanikolaou IS, Tham TC, Tringali A, van Hooft J, Williams EJ. Papillary cannulation and sphincterotomy techniques at ERCP: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2016 Jul;48(7):657-83. doi: 10.1055/s-0042-108641. Epub 2016 Jun 14. PMID 27299638
- [Background] Vazquez-Lglesias JL, Gonzalez-Conde B, Lopez-Roses L, Estevez-Prieto E, Alonso-Aguirre P, Lancho A, Suarez F F, Nunes R. Endoscopic sphincterotomy for prevention of the recurrence of acute biliary pancreatitis in patients with gallbladder in situ: long-term follow-up of 88 patients. Surg Endosc. 2004 Oct;18(10):1442-6. doi: 10.1007/s00464-003-9185-7. Epub 2004 Aug 26. PMID 15791366
- [Background] Uomo G, Manes G, Laccetti M, Cavallera A, Rabitti PG. Endoscopic sphincterotomy and recurrence of acute pancreatitis in gallstone patients considered unfit for surgery. Pancreas. 1997 Jan;14(1):28-31. doi: 10.1097/00006676-199701000-00005. PMID 8981504
- [Background] da Costa DW, Bouwense SA, Schepers NJ, Besselink MG, van Santvoort HC, van Brunschot S, Bakker OJ, Bollen TL, Dejong CH, van Goor H, Boermeester MA, Bruno MJ, van Eijck CH, Timmer R, Weusten BL, Consten EC, Brink MA, Spanier BWM, Bilgen EJS, Nieuwenhuijs VB, Hofker HS, Rosman C, Voorburg AM, Bosscha K, van Duijvendijk P, Gerritsen JJ, Heisterkamp J, de Hingh IH, Witteman BJ, Kruyt PM, Scheepers JJ, Molenaar IQ, Schaapherder AF, Manusama ER, van der Waaij LA, van Unen J, Dijkgraaf MG, van Ramshorst B, Gooszen HG, Boerma D; Dutch Pancreatitis Study Group. Same-admission versus interval cholecystectomy for mild gallstone pancreatitis (PONCHO): a multicentre randomised controlled trial. Lancet. 2015 Sep 26;386(10000):1261-1268. doi: 10.1016/S0140-6736(15)00274-3. PMID 26460661
- [Background] Schreurs WH, Juttmann JR, Stuifbergen WN, Oostvogel HJ, van Vroonhoven TJ. Management of common bile duct stones: selective endoscopic retrograde cholangiography and endoscopic sphincterotomy: short- and long-term results. Surg Endosc. 2002 Jul;16(7):1068-72. doi: 10.1007/s00464-001-9104-8. Epub 2002 May 3. PMID 11984690
- [Background] Manes G, Paspatis G, Aabakken L, Anderloni A, Arvanitakis M, Ah-Soune P, Barthet M, Domagk D, Dumonceau JM, Gigot JF, Hritz I, Karamanolis G, Laghi A, Mariani A, Paraskeva K, Pohl J, Ponchon T, Swahn F, Ter Steege RWF, Tringali A, Vezakis A, Williams EJ, van Hooft JE. Endoscopic management of common bile duct stones: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2019 May;51(5):472-491. doi: 10.1055/a-0862-0346. Epub 2019 Apr 3. PMID 30943551